CLINICAL TRIAL: NCT03840746
Title: 6 Week Feeding Study of Interactions Between Fibre and Polyphenols Sources on Colonic Phenolic Acid Production and Biomarkers of Health
Brief Title: Interactions Between Fibre and Polyphenols on Colonic Phenolic Acid Production and Biomarkers of Health ( 6 Weeks)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Scottish Universities Environmental Research Centre (Other)
Responsible Party: Principal Investigator, Christine Edwards, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BB/M027724/1-3
Record Dates: First submitted 2019-01-18; First posted 2019-02-15 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: self-reported healthy adults; age 40-70; BMI > 25
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Intervention Model Description: This intervention study will be carried out using a parallel design, with three arms (foods containing polyphenol+NDC, foods with polyphenol alone, and habitual diet control)
Who Masked: Participant, Investigator
Masking Description: soups in plain tins and labelled A or B. Code held by person not part of study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Habitual diet (No Intervention): participants remain on their habitual diet
- Tomato, onion and lovage soup (TOL) (Experimental): One tin of soup containing Tomato onion and lovage daily for 6 weeks
  Interventions: Other: Tomato, onion and lovage soup (TOL)
- TOL soup with inulin (Experimental): One tin of Tomato, onion and lovage soup with added inulin for 6 weeks
  Interventions: Other: TOL soup with inulin

INTERVENTIONS:
Other: Tomato, onion and lovage soup (TOL) — Soup
  Arms: Tomato, onion and lovage soup (TOL)
Other: TOL soup with inulin — Soup
  Arms: TOL soup with inulin

SUMMARY:
The investigators have studied the acute interactions of polyphenols and NDC in a single meal in a human study containing tomatoes, lovage & onions, with and without inulin. The investigators now wish to study the longer-term interactions of these foods over 6 weeks as well as their impact on biomarkers of human health, the gut microbiome, human proteome and markers of risk of chronic disease. This may allow better targeted evaluation of foods which influence health through the gut microbiome.

DETAILED DESCRIPTION:
Polyphenol rich plant foods have been associated with several health benefits but their bioavailability is generally low. The majority of plant polyphenols are poorly absorbed in the small intestine and enter the colon where the colonic microbiota metabolise them to release a range of phenolic acids, which are now thought to be the main bioactive components related to the reduction in disease risk. Very little is known about the impact of other constituents of the diet on the metabolism and bacterial catabolism of these polyphenols.

Colonic bacteria are key agents in the release of the bioactive molecules from polyphenols but also ferment non-digestible carbohydrates (NDC) such as inulin to short chain fatty acids. It is likely that there are key interactions in the colonic bacterial metabolism of NDC and phenolics. The investigators hypothesize that combination of polyphenolics (in onions, tomatoes and lovage) with inulin (NDC) will increase the urinary output of bioactive phenolic acids over a 6 week feeding trial and impact on biomarkers of cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* BMI>=25
* Not on antibiotics within 3 months of starting of study
* No medication likely to influence gut function, colonic bacterial activity.

Exclusion Criteria:

* Antibiotics
* Pregnancy
* lactation

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of total amount of phenolic acids (umoles/24 hours) in urine (3 wk) | 3 weeks
  Profile and amounts of phenolic acids in urine derived from the colonic bacterial metabolism of polyphenols
Change from baseline of total amount of phenolic acids (umoles/24 hours) in urine (6 wk) | 6 weeks
  Profile and amounts of phenolic acids in urine derived from the colonic bacterial metabolism of polyphenols

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT03840746/Prot_SAP_000.pdf